CLINICAL TRIAL: NCT00977197
Title: A Placebo-Controlled Trial of Pregabalin (Lyrica) for Irritable Bowel Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Yuri A. Saito Loftus, PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 09-004404
Record Dates: First submitted 2009-09-11; First posted 2009-09-15 (Estimated); Results first posted 2016-07-14 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-09

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pregabalin (Active Comparator): Subjects randomized to this arm will receive the following dosage:
  75 mg (one tablet) twice a day for three days, increasing to 150 mg (2 tablets) twice a day for three days, escalating to 225 mg (three tablets) twice a day, through week 12, day 1. Days 2-4 of week 12, participants will begin tapering and will receive 150 mg (two tablets) two times a day and then days 5-7, participants will receive 75 mg two times a day for the duration of the study.
  Interventions: Drug: Pregabalin
- Placebo (Placebo Comparator): Subjects randomized to this arm will receive placebo matching the study drug.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pregabalin — Dose: 75 mg twice a day for three days, increasing to 150 mg (2 tablets) twice a day for three days, escalating to 225 mg (three tablets) twice a day, through week 12, day 1. Days 2-4 of week 12, participants will begin tapering and will receive 150 mg (two tablets) two times a day and then days 5-7, participants will receive 75 mg two times a day for the duration of the study.
  Other Names: Lyrica
  Arms: Pregabalin
Drug: Placebo — A matching placebo will be administered twice a day
  Arms: Placebo

SUMMARY:
This study is being done to see if Lyrica helps people with irritable bowel syndrome.

DETAILED DESCRIPTION:
Lyrica is the trade name for pregabalin, which was first approved by the FDA in June 2005 and has been available through prescription since fall 2005, and is marketed by Pfizer. Lyrica is known to have clinical efficacy treating pain disorders including irritable bowel syndrome-related conditions such as fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of Irritable Bowel Syndrome (IBS)
* Experience pain with relief with defecation
* 50/100 or greater of pain or discomfort scores during the two-week baseline period
* At least three pain attacks in a month, with at least three episodes of pain intensity equal to or exceeding 50/100
* U.S. resident
* English-speaking (able to provide consent and complete questionnaires)
* Able to participate in all aspects of the study

Exclusion Criteria:

* Known alternative/concurrent gastrointestinal diagnosis (e.g. Crohn's disease, ulcerative colitis, microscopic colitis, active celiac sprue, chronic pancreatitis or pancreatic insufficiency, scleroderma, chronic intestinal pseudo-obstruction, bacterial overgrowth, recent (<6 months) intestinal bacterial/protozoal/ parasitic infections, HIV, active pelvic floor dysfunction, paraplegia or quadriplegia);
* Current symptoms of severe depression, as measured by Hospital Anxiety and Depression Scale (HADS) score (greater or less than 15);
* Mental retardation or any condition requiring a legal guardian;
* Current or past history of psychotic disorder (schizophrenia, bipolar disorder)
* Recent or current use (within past 30 days) of drugs that interact with Pregabalin:
* Rosiglitazone (Avandia) or Pioglitazone (Actos)
* Narcotic anti-pain medications (e.g. oxycodone, morphine)
* Anti-anxiety medications (e.g. lorazepam, alprazolam, diazepam)
* Unable to withdraw medications at least 72 hours prior to the study, because we will evaluate patient's response to pregabalin therapy for relief of IBS-associated pain and disturbed sleep.

  1. Non-narcotic anti-pain medications (e.g. nonsteroidal antiinflammatory drug (NSAIDs), ultram, neurontin, etc.)
  2. Mexiletine, steroids, dextromethorphan.
  3. Insomnia medications (e.g. benzodiazepines, zolpidem, diphenhydramine, melatonin, etc.)
* Planned surgery (especially transplant) or anesthesia exposure during trial
* Are pregnant, lactating, likely to become pregnant during medication phase and not willing to use a reliable form of contraception (barrier contraceptives, diaphragm, injections, intrauterine device, surgical sterilization, or abstinence)
* Recent or current use (within 30 days) of Pregabalin
* Known allergy to Pregabalin
* Significant acute or chronic progressive neurologic, hepatic, renal, cardiovascular, respiratory or metabolic disease
* Recent history of alcohol or substance dependence use or abuse
* Another household member or relative participating in the study
* Professional drivers or operators of heavy machinery
* Major cardiovascular events in the last 6 months
* Use of IBS-specific drugs such as tegaserod (Zelnorm) and Lotronex (Alosetron) (within 30 days)
* Participation in another clinical trial (within 30 days)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2010-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yuri A Saito Loftus, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - Mayo Clinic Health System - Franciscan Healthcare in La Crosse, La Crosse, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Pregabalin: Subjects randomized to this arm will receive the following dosage:
  75 mg (one tablet) twice a day for three days, increasing to 150 mg (2 tablets) twice a day for three days, escalating to 225 mg (three tablets) twice a day, through week 12, day 1. Days 2-4 of week 12, participants will begin tapering and will receive 150 mg (two tablets) two times a day and then days 5-7, participants will receive 75 mg two times a day for the duration of the study.
  Pregabalin: Dose: 75 mg twice a day for three days, increasing to 150 mg (2 tablets) twice a day for three days, escalating to 225 mg (three tablets) twice a day, through week 12, day 1. Days 2-4 of week 12, participants will begin tapering and will receive 150 mg (two tablets) two times a day and then days 5-7, participants will receive 75 mg two times a day for the duration of the study.
Period: Overall Study
Arm/Group | Pregabalin | Placebo
Started | 41 | 44
Completed | 32 | 35
Not Completed | 9 | 9
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Adverse Event | 3 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Lost to Follow-up | 1 | 3
Not completed — Nonadherence | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregabalin | Placebo | Total
Number analyzed (Participants) | 41 | 44 | 85
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 2 | 3
  Between 18 and 65 years | 38 | 40 | 78
  >=65 years | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 37 | 73
  Male | 5 | 7 | 12
Region of Enrollment [Number; unit: participants]
  United States | 41 | 44 | 85
Number of Subjects with Fibromyalgia at Baseline [Number; unit: participants]
  Fibromyalgia - No | 31 | 37 | 68
  Fibromyalgia - Yes | 10 | 7 | 17

OUTCOME MEASURES:

1. Primary Outcome: Mean Pain Bowel Symptom Scale (BSS) Score Over Last 4 Weeks of Study (Weeks 9-12)
Description: The Bowel Symptom Scale (BSS) consists of 5 questions, each with a 100 mm long Visual Analog Scale (VAS). The questions are regarding pain, bloating, constipation, diarrhea, and overall severity of Irritable Bowel Syndrome (IBS) symptoms. The VAS does not have any pre-set marks between the extremes of 0 for not present and 100 mm for very severe symptoms. The investigator measures the mark made by the participant in mm and records this for the value.
Time Frame: weeks 9-12
Population: Intent to treat analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 41 | 44
units on a scale | 25.3 (16.0) | 42.0 (26.6)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.008, ANCOVA; Intent to Treat analysis; adjusted for age and gender

2. Secondary Outcome: Mean Overall Severity of Irritable Bowel Syndrome (IBS) Symptoms BSS Score Last 4 Weeks of the Study (Weeks 9-12)
Description: as for outcome 1
Time Frame: weeks 9-12
Population: The analysis population is different than the participant flow because some subjects didn't return for a follow-up visit, or didn't complete the questionnaire.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 29 | 35
units on a scale | 26.5 (15.2) | 42.2 (25.7)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.009, ANCOVA; Intent to Treat analysis; adjusted for age and gender

3. Secondary Outcome: Mean Constipation BSS Score Over Last 4 Weeks of Study (Weeks 9-12)
Description: as for outcome 1
Time Frame: Weeks 9-12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 29 | 35
units on a scale | 25.8 (26.8) | 22.4 (24.8)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.389, ANCOVA; Intent to Treat analysis; adjusted for age and gender; rank scale

4. Secondary Outcome: Mean Diarrhea BSS Score Over the Last 4 Weeks of the Study (Weeks 9-12)
Description: as for outcome 1
Time Frame: Weeks 9-12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 29 | 35
units on a scale | 16.9 (18.4) | 31.8 (25.8)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.049, ANCOVA; Intent to Treat analysis; adjusted for age and gender, rank scale

5. Secondary Outcome: Mean Bloating BSS Score Over the Last 4 Weeks of the Study (Weeks 9-12)
Description: as for outcome 1
Time Frame: Weeks 9-12)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 29 | 35
units on a scale | 29.3 (23.3) | 43.6 (29.0)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.044, ANCOVA; Intent to Treat analysis; adjusted for age and gender

6. Secondary Outcome: Number of Subjects With Adequate Relief of IBS Symptoms at Least 50% of the Last 4 Weeks of Therapy
Description: One of the weekly questions asked of subjects was, "Did you have adequate relief of your IBS symptoms over the last week?" Possible answers were Yes or No.
Time Frame: Weeks 9-12
Population: Intent to treat analysis
Measure: Number; unit: participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 41 | 44
participants
  Adequate Relief (Yes) | 19 | 16
  Inadequate Relief (No) | 22 | 28
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.350, Chi-squared — Intent to treat analysis, not adjusted for age and gender

7. Secondary Outcome: Mean Pain BSS Score at Week 12
Description: as for outcome 1
Time Frame: Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 29 | 34
units on a scale | 26.1 (18.8) | 43.3 (30)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.020, ANCOVA; Intent to Treat analysis; adjusted for age and gender, rank scale

8. Secondary Outcome: Mean Overall Severity BSS Score at Week 12
Description: as for outcome 1
Time Frame: Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 29 | 34
units on a scale | 28.5 (20.2) | 44.2 (28.8)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.024, ANCOVA; Intent to Treat analysis; adjusted for age and gender

9. Secondary Outcome: Mean Constipation BSS Score at Week 12
Description: as for outcome 1
Time Frame: Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 29 | 34
units on a scale | 26.1 (30.4) | 23.6 (26.7)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.417, ANCOVA; Intent to Treat analysis; adjusted for age and gender, rank scale

10. Secondary Outcome: Mean Diarrhea BSS Score at Week 12
Description: as for outcome 1
Time Frame: Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 29 | 34
units on a scale | 15.6 (19.8) | 34.4 (29.7)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.030, ANCOVA — Intent to Treat analysis; adjusted for age and gender, rank scale

11. Secondary Outcome: Mean Bloating BSS Score at Week 12
Description: as for outcome 1
Time Frame: Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 29 | 34
units on a scale | 26.3 (24.4) | 45.0 (32.0)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.016, ANCOVA; Intent to Treat analysis; adjusted for age and gender

12. Secondary Outcome: Number of Subjects With Greater Than or Equal to a 30 Point Change in Pain BSS Score
Description: as for outcome 1
Time Frame: baseline, week 12
Population: Intent to Treat analysis
Measure: Number; unit: participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 41 | 44
participants
  Yes, >= 30 point change | 26 | 20
  No, >= 30 point change | 15 | 24
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.097, Chi-squared — Intent to Treat analysis; not adjusted for age and gender

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Pregabalin | Placebo
Serious Adverse Events (participants affected / at risk) | 1/41 | 0/44
Other Adverse Events (participants affected / at risk) | 28/41 | 24/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pregabalin (N=41) | Placebo (N=44)
External Trauma (Social circumstances) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pregabalin (N=41) | Placebo (N=44)
Insomnia (General disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 6 (7) | 7 (11)
Tired (General disorders) | 6 (9) | 5 (5)
Pain in lower chest (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Cramping right side (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 6 (6) | 5 (5)
Dizzy (Nervous system disorders) | 13 (20) | 2 (2)
Blurred Vision (Eye disorders) | 6 (6) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 13 (15) | 13 (17)
Bloating (Gastrointestinal disorders) | 4 (4) | 5 (6)
Migraine (Nervous system disorders) | 2 (2) | 1 (1)
Upset stomach (Gastrointestinal disorders) | 4 (7) | 1 (1)
Flu like symptoms (Infections and infestations) | 1 (1) | 1 (1)
Heart racing (Cardiac disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 9 (11) | 4 (4)
Mucus in bowel movement (Gastrointestinal disorders) | 2 (4) | 0 (0)
Weight gain (General disorders) | 1 (1) | 0 (0)
Restless at night (General disorders) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (6) | 2 (2)
Body aches (General disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Abdominal gas (Gastrointestinal disorders) | 4 (4) | 4 (5)
Stress (General disorders) | 1 (1) | 2 (2)
Feeling of being high or tipsy (Nervous system disorders) | 4 (6) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Paresthesia (tingling) of the fingers (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Fullness in the abdomen (Gastrointestinal disorders) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Itch (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0)
Respiratory symptoms (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Leg cramps (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Burping (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dry eyes (Eye disorders) | 1 (2) | 1 (1)
More bowel movements than usual (Gastrointestinal disorders) | 2 (2) | 2 (2)
Loss of appetite (Gastrointestinal disorders) | 0 (0) | 1 (1)
No libido (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pain in upper right chest (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Excessive thirst (Gastrointestinal disorders) | 0 (0) | 1 (1)
Blood pressure increased (Cardiac disorders) | 0 (0) | 1 (1)
Muscle pain rib cage right side (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain over all body (General disorders) | 0 (0) | 1 (1)
Pain lower left side (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fingers swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Urgency to defecate (Gastrointestinal disorders) | 0 (0) | 1 (1)
Foot peripheral edema (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Gout in arches of feet (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bladder infection (Infections and infestations) | 0 (0) | 1 (1)
Increased hunger (General disorders) | 0 (0) | 1 (1)
Muscle twitching in upper back (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Change in appearance of stool (Gastrointestinal disorders) | 0 (0) | 3 (3)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Vivid dreams (General disorders) | 0 (0) | 1 (1)
Nerve pain down arms and legs (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Loss of nails (General disorders) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes